CLINICAL TRIAL: NCT03037489
Title: An Open-Label, One-Arm Phase II Extension Study to Evaluate Safety and Tolerability of MIV-711 in Patients With Knee Joint Osteoarthritis
Brief Title: A Study to Evaluate Safety and Tolerability of MIV-711 in Osteoarthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIV-711-202
Record Dates: First submitted 2016-12-22; First posted 2017-01-31 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — MIV-711

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MIV-711 (Experimental): MIV-711 for a total of 26 weeks
  Interventions: Drug: MIV-711

INTERVENTIONS:
Drug: MIV-711 — MIV-711 administered orally once daily

SUMMARY:
This is a multicentre, open-label, one-arm Phase II extension study to evaluate the safety and tolerability of MIV-711 in patients with knee joint osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

- Previously enrolled in the MIV-711-201 study including completion of Visit 8 either by

* Receiving MIV-711 200 mg and had non-significant clinical worsening on the primary endpoint as defined by a Numeric Rating Scale (NRS) increase of ≤2 OR by
* Receiving placebo and had a clinically significant worsening on the primary endpoint as defined by a NRS increase of ≥2

Exclusion Criteria:

* The presence of any inflammatory arthritis
* Any generalized pain condition that may interfere with the evaluation of the target knee pain (e.g., fibromyalgia) as judged by the investigator.
* Any clinically severe or significant uncontrolled concurrent illness, which, in the opinion of the Investigator, would impair ability to give informed consent or take part in or complete this clinical study.
* Known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Conaghan, Professor, Principal Investigator — Leeds Institute of Rheumatic and Musculoskeletal Medicine
Locations (4):
- MC Comac Medical, Sofia, Bulgaria
- LCC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- PAREXEL Berlin Early Phase Clinical Unit, Berlin, Germany
- LCC ARENSIA Exploratory Medicine, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Study Group A was recruited from patients treated with 200 mg MIV-711 once daily in Study MIV-711-201 (NCT02705625) and whose symptoms did not clinically significantly deteriorate as defined by an increase in the Numeric Rating Scale (NRS) of ≤2 compared to baseline. Patients in Study Group A continued the same dosing with 200 mg MIV-711 once daily for 26 additional weeks.
- Group B: Study Group B was recruited from patients receiving placebo in Study MIV-711-201 (NCT02705625) having experienced a clinical worsening as defined by an increase in NRS of ≥2 versus baseline. Patients in Study Group B were treated with 200 mg MIV-711 once daily for the next 26 weeks.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 46 | 4
Completed | 39 | 4
Not Completed | 7 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Study Group A was recruited from patients treated with 200 mg MIV-711 once daily in Study MIV-711-201 and whose symptoms did not clinically significantly deteriorate as defined by an increase in the NRS of ≤2 compared to baseline. Patients in Study Group A continued the same dosing with 200 mg MIV-711 once daily for 26 additional weeks.
- Group B: Study Group B was recruited from patients receiving placebo in Study MIV-711-201 having experienced a clinical worsening as defined by an increase in NRS of ≥2 versus baseline. Patients in Study Group B were treated with 200 mg MIV-711 once daily for the next 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 46 | 4 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 2 | 32
  >=65 years | 16 | 2 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.52) | 65.5 (5.51) | 61.8 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 3 | 34
  Male | 15 | 1 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 46 | 4 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Moldova | 21 | 3 | 24
  Georgia | 3 | 0 | 3
  Bulgaria | 9 | 0 | 9
  Germany | 13 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of MIV-711 in Osteoarthritis (OA) Patients
Description: 1. Number of Participants with Treatment Emergent Adverse Events (TEAEs)
  2. Number of Participants with Serious Adverse Events (SAEs)
  3. Number of Participants with TEAEs related to treatment
  4. Number of Participants with mild TEAEs
  5. Number of Participants with moderate TEAEs
  6. Number of Participants with severe TEAEs
  7. Number of Participants with TEAEs leading to early discontinuation
Time Frame: Group A: 0-56 weeks; Group B: 0-30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 46 | 4
Participants
  TEAEs | 21 | 2
  SAEs | 2 | 0
  Related TEAEs | 1 | 0
  Mild TEAEs | 6 | 1
  Moderate TEAEs | 14 | 1
  Severe TEAEs | 1 | 0
  TEAEs leading to early discontinuation | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing the Informed Consent Form to the Follow up visit (4 weeks after end of treatment), up to 56 weeks.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/46 | 0/4
Other Adverse Events (participants affected / at risk) | 13/46 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=46) | Group B (N=4)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=46) | Group B (N=4)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT03037489/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03037489/SAP_001.pdf